CLINICAL TRIAL: NCT04160728
Title: Occupational Heat Stress on Workers' Productivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 7. Workers' heat stress
Record Dates: First submitted 2019-11-07; First posted 2019-11-13 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Risk of Heat Stress
Keywords: heat stress; heat strain; productivity; labor; occupation; work; thermal
MeSH Terms: conditions — Heat Stress Disorders | interventions — Commerce

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Work/ rest scenario (Experimental): For every hour of work, the participants were asked to take 3-10 minutes break in the shade.
  Interventions: Other: Work/ rest scenario
- Hydration scenario (Experimental): Participants were asked to consume at least 750ml of water or ice-slushies for every hour of work.
  Interventions: Other: Hydration scenario
- Clothing scenario (Experimental): Participants were asked to wear different types of clothing during the work shift i.e. ventilated garments, white breathable coveralls, clothing with water submerged parts.
  Interventions: Other: Clothing scenario
- "E-carts" scenario (Experimental): Participants that were involved in manual labor by carrying heavy weights were provided with "e-carts" (automated carrying vehicles)
  Interventions: Other: "E-carts" scenario
- Business as usual scenario (Sham Comparator): No interference with the usual work day of the participants.
  Interventions: Other: Business as usual scenario
- Sham evaluation (Sham Comparator): Participants were monitored during a usual day of work shift while sham measurements were recorded in order for them to get familiarized with the study environment.
  Interventions: Other: Sham evaluation

INTERVENTIONS:
Other: Work/ rest scenario — For every hour of work, the participants were asked to take 3-10 minutes break in the shade.
  Arms: Work/ rest scenario
Other: Hydration scenario — Participants were asked to consume at least 750ml of water or ice-slushies for every hour of work
  Arms: Hydration scenario
Other: Clothing scenario — Participants were asked to wear different types of clothing during the work shift i.e. ventilated garments, white breathable coveralls, clothing with water submerged parts
  Arms: Clothing scenario
Other: "E-carts" scenario — Participants that were involved in manual labor by carrying heavy weights were provided with "e-carts" (automated carrying vehicles)
  Arms: "E-carts" scenario
Other: Business as usual scenario — No interference with the usual work day of the participants
  Arms: Business as usual scenario
Other: Sham evaluation — Participants were monitored during a usual day of work shift while sham measurements were recorded in order for them to get familiarized with the study environment
  Arms: Sham evaluation

SUMMARY:
Workplace heat exposure affects billions of people during their everyday work activities. Occupational heat stress impairs workers' health and capacity to perform manual labour. Therefore, the aim of this study was to observe the heat strain experienced by workers in occupational settings and test different strategies to mitigate it during actual work shifts in agriculture, manufacture, tourism, construction, and other services.

DETAILED DESCRIPTION:
The participants followed the study protocol which included, one work shift of sham measurements, one work shift business as usual and four (4) different scenarios (interventions) on different work shifts. Apart from the sham measurements the rest of the scenarios were tested in a random order for different participants.

1. Work/ rest scenario: The participants were asked to take planned breaks in the shade during their work shift. The amount of breaks taken ranged between 3 and 10 minutes every hour depending on the current work duties of the employees.
2. Hydration scenario: The participants were advised (not forced) to drink minimum of 750 ml of water or ice - slushies, every hour during their work shift.
3. Clothing scenario: The participants were randomly provided with different types of clothing, i.e. white breathable coveralls, ventilated garments and breathable uniform with water submerging parts, to wear during their work shift.
4. Assisted labor: The participants in agriculture, that were carrying heavy weights were provided with "e-carts" (automated carrying vehicles), during their work shift.

Baseline data [self-reported age; body stature (Seca 213; seca GmbH & Co. KG; Hamburg, Germany) and body mass (BC1000, Tanita corporation, Tokyo, Japan)] were collected one day prior to the measurements. Medical history of all the participants was recorded. During the field study, continuous heart rate, core temperature and mean skin temperature data were collected using wireless heart rate monitors (Polar Team2. Polar Electro Oy, Kempele, Finland), telemetric capsules (BodyCap, Caen, France), and wireless thermistors (iButtons type DS1921H, Maxim/Dallas Semiconductor Corp., USA), respectively. Skin temperature data were collected from four sites (chest, arm, thigh, and leg) and were expressed as mean skin temperature according to the formula of Ramanathan (Tsk = [0.3(chest + arm) + 0.2(thigh + leg)]). Furthermore, continuous environmental data [air temperature (°C), globe temperature (°C), relative humidity (%), and air velocity (m/s)] were collected using a portable weather station (Kestrel 5400FW, Nielsen-Kellerman, Pennsylvania, USA). Urine samples were collected at the start and the end of the work shift to evaluate the hydration status of each worker. Urine specific gravity was assessed for each urine sample using a refractometer (PAL-10S, ATAGO CO., LTD., Fukaya, Saitama Prefecture, Japan) and was classified as either hydrated (< 1.020) or dehydrated (≥ 1.020). In addition, urine colour was assessed using a urine color scale. Questionnaires were used to assess workers' perception on exertion (Borg scale), thermal comfort/sensation, humidity comfort/sensation, radiation comfort/sensation, wind speed comfort/sensation, skin wetness, sleepiness, physical demands of the workload. The Heat Strain Score Index (HSSI) was used to assess the perceived heat strain of the workers.

Video cameras installed in close proximity (about 40m) to the workers were used to assessed workers labour effort. Video recordings were analyzed on a second by second basis using time-motion analysis method. Importantly, when video cameras were not feasible to be installed real-time task analysis was used to examine workers capacity for manual labour. For that reason, an android-based application (FAME_TASK App) was used to record the tasks of the workers on a second by second basis. The App was continuously monitoring the work time spent on irregular work breaks (unplanned breaks), the duration of uninterrupted work and the time spent as lunch time or other breaks provided by management (planned breaks). The unplanned break was divided into two categories: the breaks during which the workers decided to rest in the shade (unplanned break under the shade) and the breaks during which the workers chose to stay under the sun (unplanned break under the sun). Also, the uninterrupted work was divided into nine categories: work in an outdoor environment with a low metabolic rate; work in an outdoor environment with a moderate metabolic rate; work in an outdoor environment with a high metabolic rate; work in a mixed (outdoor and indoor) environment with a low metabolic rate; work in a mixed (outdoor and indoor) environment with a moderate metabolic rate; work in a mixed (outdoor and indoor) environment with a high metabolic rate; work in an indoor environment with a low metabolic rate; work in an indoor environment with a moderate metabolic rate; work in an indoor environment with a high metabolic rate. The labor effort (i.e., low / moderate / high metabolic rate) was defined according to the ISO 8996:1994 as low, moderate and high metabolic rate. Based on these definitions, the recorded tasks were fourteen. During the work-shift, a researcher was following each worker, monitoring them with the FAME_TASK App, until they end of their work shift.

ELIGIBILITY:
Inclusion Criteria:

* Workers in the industries of agriculture, construction, manufacture, , tourism, or other services

Exclusion Criteria:

* Workers under the age of 18 or non-experienced workers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
Heart rate | 12-hour workshift
  Heart rate data were continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Mean skin temperature | 12-hour workshift
  Temperature at the skin surface area was continuously monitored using iButton sensors (type DS1921 H, Maxim/Dallas Semiconductor Corp., USA)
Core body temperature | 12-hour workshift
  Core body temperature was assessed throughout the entire work shift using telemetric capsules (e-Celsius, BodyCap, Caen, France) that was given to the workers to ingest prior to their work shift
Urine specific gravity to assess the hydration status | Pre and post the 12-hour workshift
  Urine was obtained from the participants pre and post the 12-hour work shift. Urine specific gravity (single assessment-no units) was assessed using a refractometer (PAL-10S, ATAGO CO., LTD., Fukaya, Saitama Prefecture, Japan). Urine color was assessed using a urine color scale
Labour effort | 12-hour workshift
  Actual time (single assessment-hours) of working effort and break time during the 12-hour work shift. They were assessed by time-motion analysis (video) or real time task analysis (surveillance) on a second by second basis
Thermal comfort | At baseline, every two hours up until the end of the 12-hour workshift
  Thermal comfort was assessed via the thermal comfort scale (1 = comfortable; 5 = extremely uncomfortable).
Thermal sensation | At baseline, every two hours up until the end of the 12-hour workshift
  Thermal sensation was assessed via the thermal sensation scale (-3 = cold; +3 = hot)
Perceived exertion | At baseline, every two hours up until the end of the 12-hour workshift
  Perceived exertion was assessed via the Borg 20th Scale (6 = no exertion at all; 20 = maximal exertion)
Heat Strain Score Index | At the end of the 12-hour work shift
  Heat Strain Score Index was assessed via the 18-question Heat Strain Score Index questionnaire that assess the heat and physiological strain

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Flouris, Principal Investigator — andreasflouris@gmail.com
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ioannou LG, Tsoutsoubi L, Mantzios K, Gkikas G, Agaliotis G, Koutedakis Y, Garcia-Leon D, Havenith G, Liang J, Arkolakis C, Glaser J, Kenny GP, Mekjavic IB, Nybo L, Flouris AD. The Impact of Workplace Heat and Cold on Work Time Loss. J Occup Environ Med. 2025 Jun 1;67(6):393-399. doi: 10.1097/JOM.0000000000003332. Epub 2025 Feb 7. PMID 39965897